CLINICAL TRIAL: NCT05064202
Title: Use of mechaNical Left ventricuLar unlOading in Acute decompensateD Heart Failure Complicated by Cardiogenic Shock - the UNLOAD HF-CS Trial.
Brief Title: Unloading in Heart Failure Cardiogenic Shock
Acronym: UNLOAD HF-CS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Principal Investigator, Alexander Nap, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL84199.018.23
Record Dates: First submitted 2021-08-26; First posted 2021-10-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cardiogenic Shock
Keywords: Unloading; Acute Decompensated Heart Failure; Cardiogenic Shock; temporary Mechanical Circulatory Support (tMCS); Inotropes
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Impella 5.5 (Experimental): ADHF-CS patients who are in the experimental arm will be treated with an Impella 5.5 (+/- standard of care)
  Interventions: Device: Impella 5.5
- Standard of care (Other): ADHF-CS patients who are in the control arm will be treated with escalating doses of inotropes (standard of care)
  Interventions: Drug: Inotropes

INTERVENTIONS:
Device: Impella 5.5 — temporary Mechanical Circulatory Support (tMCS)
  Arms: Impella 5.5
Drug: Inotropes — Enoximone, Dobutamine, Dopamine, Milrinone
  Arms: Standard of care

SUMMARY:
The purpose of this research study is to evaluate whether timely and aggressive temporary Mechanical Circulatory Support (tMCS) through the Impella 5.5® in patients with acute decompensated heart failure complicated by cardiogenic shock (ADHF-CS) has the potential to reduce the HF-CS related clinical events compared to the current standard of care.

DETAILED DESCRIPTION:
To demonstrate the efficacy of timely temporary mechanical left ventricular unloading with the Impella 5.5® assist device in patients with acute decompensated heart failure complicated by cardiogenic shock (ADHF-CS) vs. current standard of (pharmacological) care

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of HFrEF according to ESC HF guidelines (LVEF ≤ 35%) 2. Signs of (persistent) congestion (elevated CVP, edema, rales, ascites, pleural effusion) 3. Evidence of CS with presence of at least 2 of the 3 following:

1. Hypotension

   1. systolic blood pressure <90 mmHg for at least 30 min OR
   2. mean arterial pressure <60 mmHg for at least 30 min
2. Hypoperfusion

   1. lactate > 2.0 mmol/L (two consecutive values > 2 mmol/L with at least 30 min between samples, with non-decreasing trend on if on (steady doses of) inotropes and/or vasopressors)
   2. amino-L-transferase >200 U/L (two consecutive values > 200 Ul/L with at least 30 min between samples, with non-decreasing trend if on (steady doses of) inotropes and/or vasopressors)
   3. creatinine rise ≥ 0.3 mg/dl/24h ( 26,53 μmol/L)
   4. oliguria (≤ 0,5 ml/kg/h, ≤ 720 ml/24 h)
3. Inotropes/vasoactives (use of)

Exclusion Criteria:

1. Contraindications for Impella 5.5
2. Severe concomitant RV failure
3. Grade IV mitral regurgitation eligible for surgical treatment
4. Dialysis for end-stage renal failure
5. Acute coronary syndrome (type 1, AMI)
6. Bradycardia and AV blocks necessitating pacemaker implantation
7. HD parameters and biochemistry alterations as specifically defined for SCAI CS E
8. Combined cardiorespiratory failure
9. Resuscitated (OHCA/PEA)
10. History of CVA or TIA within previous 90 days
11. History of acute myocardial infarction within previous 30 days
12. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombo-cytopenia), any recent GU or GI bleed, or will refuse blood transfusions
13. Inflammatory
14. Active systemic infections
15. Acute myocarditis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality, renal replacement therapy and rehospitalization or urgent visit for heart failure (Efficacy - Primary Combined Clinical Endpoint) | baseline to 90 days
  Number of patients suffering from any of: all-cause death, renal replacement therapy and rehospitalization or urgent hospital visit for heart failure up to 90 days

SECONDARY OUTCOMES:
In-hospital mortality (Efficacy - Secondary Endpoint) | baseline to 28 days
  Number of patients suffering from cardiac death and non-cardiac death and undetermined death during hospitalisation
In-hospital Worsening Heart Failure (Efficacy - Secondary Endpoint) | baseline to 28 days
  Number of patients with progression to SCAI CS stage D OR E (depending on stage directly after randomization)
Cardiac mortality (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that died of any cause at 90 days and 1 year
All-cause mortality (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that died of any cause at 90 days and 1 year
Mechanical ventillation (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that were mechanically ventilated during hospitalization, up to day 90 and 1 year
Renal replacement therapy (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that received renal replacement therapy during hospitalization, up to day 90 and 1 year
Hospitalization or urgent hospital visit for heart failure (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that were hospitalized or had an urgent hospital visit for heart failure up to day 30, 60 and 1 year
Urgent / rescue MCS implantation (permanent) (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that received a permanent MCS device implantation up to day 90 and 1 year
Hospitalization time (Efficacy - Secondary Endpoint) | baseline to 28 days
  Lenght of index hospitalization for HF-CS in days
Vasoactive Inotropic Score (maximal) (Efficacy - Secondary Endpoint) | baseline to 28 days
  Maximal VIS during hospitalization
LVAD / Heart transplantation (Efficacy - Secondary Endpoint) | baseline to 1 year
  Number of patients that received heart treplacement therapy up to discharge, 90 days and 1 year
KCCQ-12 (Efficacy - Secondary Endpoint) | 90 days, 1 year
  Average KCCQ-12 at 90 days and 1 year
Stroke or TIA (Safety - Secondary Endpoint) | baseline to 28 days
  Number of patients that developed a stroke or TIA up to discharge
Major Bleeding (Safety - Secondary Endpoint) | baseline to 28 days
  Number of patients that developed a major bleed up to discharge
Major vascular events (Safety - Secondary Endpoint) | baseline to 28 days
  Number of patients that developed a major vascular event up to discharge
Extremity ischemia (Safety - Secondary Endpoint) | baseline to 28 days
  Number of patients that developed limb ischemia up to discharge
Hemolysis (Safety - Secondary Endpoint) | baseline to 28 days
  Number of patients diagnosed with hemolysis up to discharge
Insertion site infection (Safety - Secondary Endpoint) | baseline to 28 days
  Number of patients that developed an infection at the insertion site up to discharge
Aortic valve injury (Safety - Secondary Endpoint) | baseline to 90 days
  Number of patients that developed aortic valve insufficiency (by echo) up to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Nap, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (5):
- Netherlands (5):
  - Academical Medical Center (AMC), Amsterdam
  - VU University Medical Center (VUMC), Amsterdam
  - Univerity Medical Center Groningen (UMCG), Groningen
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - University Medical Center Utrecht (UMCU), Utrecht

IPD SHARING:
Plan to Share IPD: No